CLINICAL TRIAL: NCT04629300
Title: Randomized Trial of a Supportive Care Mobile Application to Improve Symptoms, Coping, and Quality of Life in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Supportive Care Mobile Application for Patients With NSCLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-398
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer; Quality of Life; Coping Skills
Keywords: Non Small Cell Lung Cancer; Portable Electronic Applications; Quality of Life; Coping Skills
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Care Mobile Application (Experimental): Complete study questionnaires at two time points:
  * upon enrollment at baseline prior to randomization
  * approximately 12 weeks after the baseline assessment time point.
  Participants will be provided with a study-issued tablet computer to access mobile app and receive a comprehensive tutorial and detailed instructions on how to use the app.
  Participants will have approximately 10 weeks to complete the intervention modules at self initiated pace. The app will provide prompts as reminders to complete the modules.
  Participants will receive standard oncology care. Study staff will monitor participant use of supportive care services, such as social work, psychology, psychiatry, and palliative care.
  Interventions: Behavioral: Supportive Care Mobile Application; Other: Usual Care
- Usual Care (Active Comparator): Complete study questionnaires at two time points:
  * upon enrollment at baseline prior to randomization
  * approximately 12 weeks after the baseline assessment time point.
  Participants will receive standard oncology care. Study staff will monitor participant use of supportive care services, such as social work, psychology, psychiatry, and palliative care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Supportive Care Mobile Application — Tablet computer with application providing modules on skills for managing symptoms and coping.
  Arms: Supportive Care Mobile Application
Other: Usual Care — Standard oncology care with monitoring of supportive care services usage

SUMMARY:
This research study is looking at the role of a supportive care mobile app in improving symptoms, coping skills, and quality of life in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first-time investigators are examining this supportive care mobile app intervention. The goal of this research study is to refine and examine the feasibility and benefits of a supportive care mobile app to improve symptoms, coping skills, and quality of life in patients with non-small cell lung cancer. Many people diagnosed with lung cancer experience challenging symptoms and increased stress. To help address these concerns, this study is exploring how a mobile application (app) intervention, designed specifically for people with lung cancer, can expand the availability of much needed supportive care services.

The research study procedures include:

* A supportive care mobile app consisting of six intervention modules that focus on components of wellbeing, such as physical, social, functional, and emotional wellbeing
* Questionnaires asking about demographic information (e.g., gender, ethnicity, income) and participants' experience with cancer (e.g., quality of life, symptoms)
* Data collection from participants medical records

After completing a baseline study questionnaire, participants will be randomized into two (2) study groups:

* Usual Care Group: Participants will receive standard oncology care and attend their regular clinic visits. Study staff will monitor participant use of supportive care services.
* Intervention Group: Participants will be provided with a study-issued tablet computer to access the mobile app and receive tutorial and instructions for how to use the app.

Participants will be in this research study for 12-14 weeks.

It is expected that about 120 people will take part in this research study.

The sponsors of this study are the National Comprehensive Cancer Network (NCCN) and AstraZeneca Pharmaceuticals. NCCN is a non-profit alliance of leading cancer centers across the United States, and AstraZeneca Pharmaceuticals is a global bio-pharmaceutical company. These two sponsors are together providing funding and oversight for the conduct of this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosed with unresectable Stage III or IV NSCLC in the past twelve weeks and receiving care with palliative intent (per clinician documentation in the electronic health record)
* Eastern Cooperative Oncology Group Performance Status = 0-3
* Plan to receive oncology care at one of the participating study sites
* Ability to read and respond to questions in English

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder (e.g., psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (e.g., dementia, cognitive impairment), which the treating oncology clinician reports would prohibit the ability to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Study feasibility based on rates of participant recruitment and completion of assigned study procedures | 12 weeks
  Study feasibility will be defined as ≥ 65% approach-to-enrollment rate of eligible participants and
  ≥70% completion rate of study procedures (at least four mobile app modules and assigned study questionnaires)

SECONDARY OUTCOMES:
Patient-reported acceptability and usability of the mobile application intervention on the System Usability Scale | 12 weeks
  Describe patient-reported acceptability and ease of use of the mobile application intervention based on scores from the System Usability Scale (score range: 0-100; higher scores indicate greater acceptability and ease of use)
Compare patient-reported quality of life between study groups on the Functional Assessment of Cancer Therapy-Lung Scale | 12 weeks
  Compare between study groups patient-reported quality of life based on scores from the Functional Assessment Cancer Therapy-Lung Scale at 12 weeks (score range: 0-136; higher scores indicate better quality of life)
Compare patient-reported symptoms between study groups on the MD Anderson Symptom Inventory | 12 weeks
  Compare between study groups patient-reported symptom severity and interference based on scores from the MD Anderson Symptom Inventory at 12 weeks (score range: 0-10 on the symptom severity and interference sub-scales; higher scores indicate worse symptoms)
Compare patient-reported psychological distress between study groups on the Hospital Anxiety and Depression Scale | 12 weeks
  Compare between study groups patient-reported anxiety and depression symptoms based on scores from the Hospital Anxiety and Depression Scale at 12 weeks (score range: 0-21 on the anxiety and depression sub-scales; higher scores indicate worse psychological distress)
Compare patient-reported coping between study groups on the Brief COPE Scale | 12 weeks
  Compare between study groups patient-reported coping strategies based on scores from the Brief COPE Scale at 12 weeks (score range: 2-8 on each of 14 coping sub-scales; higher scores indicate greater use of that specific coping strategy)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Greer, PHD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Dana-Farber Brigham Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Dana-Farber Brigham Cancer Center at South Shore, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Waldman LP, Centracchio JA, Jacobs JM, Petrillo LA, El-Jawahri AR, Temel JS, Greer JA. Study protocol for a randomized trial of a supportive care mobile application to improve symptoms, coping, and quality of life in patients with advanced non-small cell lung cancer. Front Psychol. 2023 Jun 22;14:1184482. doi: 10.3389/fpsyg.2023.1184482. eCollection 2023. PMID 37425161